CLINICAL TRIAL: NCT00685282
Title: The Effect of Stress on DNA Integrity and the Effect of Cognitive Behavioral Therapy on Stress and Infertility in Women Undergoing IVF Treatment.
Brief Title: The Effect of Stress on DNA Integrity and the Effect of Cognitive Behavioral Therapy on Stress and Infertility in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Eitan Lunenfeld, Head of the IVF Unit at the Soroka Medical Center, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SOR469308CTIL
Record Dates: First submitted 2008-05-25; First posted 2008-05-28 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Infertility; Stress
MeSH Terms: conditions — Infertility | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COGNITIVE BEHAVIORAL INTERVENTIONS (Other): PSYCHOLOGICAL INTERVENTIONS TO INCLUDE, RELAXATION, STRESS REDUCTION, GUIDED IMAGERY, BREATHING EXERCISES
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The intervention (CBT) will focus on teaching specific skills which are adapted for women undergoing fertility related problems. Through the sessions the participants will learn relaxation techniques such as breathing, progressive relaxation, and guided imagery. Furthermore, suggestions for making healthier choices for coping and for releasing tension will be reviewed and discussed, with an emphasis on making healthy lifestyle changes with balance and perspective rather than in a punishing or depriving way. Each session will consist of: 20 minutes of stress-reduction behavioral relaxation, 40 minutes of cognitive restructuring and 30 minutes personal tailoring of the behavioral homework between each session.

SUMMARY:
The general hypothesis of the research is that stress decreases fertility and that Cognitive Behavioral Therapy will reduce stress and increase fertility. Secondarily, we hypothesize that stress has a detrimental effect on DNA integrity and that stress reduction will reduce DNA damage in the cell.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 18-35 without children undergoing IVF treatment

Exclusion Criteria:

* undergoing treatment for a DSM-IV axis I psychiatric illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
pregnancy | two years

SECONDARY OUTCOMES:
DNA damage/ γH2AX | with in IVF cycle (2 months)
decreased stress | two months

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Lunenfeld, PHD MD, Study Chair — Soroka UMC; Julie Cwikel, PhD, Principal Investigator — Ben-Gurion University of the Negev; Orly Sarid, PhD, Principal Investigator — Ben-Gurion University of the Negev; Iris Harvardi, PhD, Principal Investigator — Soroka UMC
Locations (1):
- IVF Clinic Soroka UMC, Beersheba, Israel